CLINICAL TRIAL: NCT05335629
Title: Evaluation of the Effect of Dapagliflozin on Cardiac Remodeling in Post Myocardial Infarction Patients
Brief Title: Evaluation of the Effect of SGLT-2 Inhibitors on Cardiac Remodeling in Post Myocardial Infarction Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdallah Heshmat, Clinical pharmacy demonstrator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dapagliflozin and ST2
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Myocardial Infarction; Diabetes Mellitus, Type 2; Myocardial Remodeling, Ventricular
Keywords: Dapagliflozin; ST2; Myocardial infarction; Cardiac remodeling; T2DM
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus, Type 2; Ventricular Remodeling | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): 30 patients will receive standard of care in addition to the SGLT2 Dapagliflozin 10 mg daily for 4 Weeks
  Interventions:
  Drug: Dapagliflozin 10 mg oral tablets Standard of care: Dual antiplatelet therapy, Statin, anticoagulation therapy
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Control arm (No Intervention): 30 patients will receive standard of care (Dual antiplatelet therapy, Statin, anticoagulation therapy) for 4 weeks

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Dapagliflozin is a sodium-glucose cotransporter-2 inhibitor (SGLT2 inhibitor) which is a new class of hypoglycemic drugs, and they can block sodium-dependent glucose transporter-2 (SGLT2) located in the early proximal renal tubule to increase urinary glucose excretion and decrease the concentration of blood glucose
  Arms: Intervention arm

SUMMARY:
A prospective, randomized, controlled study will be conducted at Clinical Cardioglogy department, Ain Shams University Hospitals, assessing the efficacy and tolerability of SGLT2 inhibitors (dapagliflozin) addition on the clinical outcome and cardiac remodeling markers of post myocardial infarction (MI) diabetic patients

DETAILED DESCRIPTION:
All patients presenting to the Clinical Cardiology department, Ain Shams University Hospitals, will be assessed for eligibility as follow:

Inclusion criteria:

1. Female or male aged >18 and < 75 years
2. Diabetic post myocardial infarction patients
3. First anterior STEMI with successful TIMI-3 flow
4. STEMI within 12 hrs of onset of chest pain
5. creatine clearance ≥60 mL/min
6. HbA1c between 6.5% and 12.0%

Exclusion criteria:

1. Cardiogenic shock on admission
2. Multivessel disease on admission
3. Mechanical complications e.g. mitral regurge on admission
4. Life threatening arrhythmia on admission
5. Hemodynamic instability on admission
6. Diagnosis of Type 1 diabetes mellitus
7. History of bladder cancer or history of radiation therapy to the lower abdomen or pelvis at any time
8. Active urinary infection diagnosed by clinical symptoms of urgency and frequency + lab tests
9. Pregnant or breast-feeding patients
10. Active participation in another clinical study
11. AST or ALT >3x ULN or Total bilirubin >2.5 x ULN
12. CrCl < 60 ml/min (based on the Cockroft-Gault equation)

Eligible patients will be randomly assigned into one of 2 arms:

1. Group 1 (Healthy control) (n=10) Aged-matched healthy volunteers who do not suffer any diseases.
2. Group 2 (Control group) (n= 30): Post-MI patients who will receive standard of care for 4 Weeks
3. Group 3 (Test group) (n= 30): Post-MI patients who will receive standard of care in addition to the SGLT2 Dapagliflozin 10 mg daily for 4 Weeks

   * Dapagliflozin will be administered immediately at time of PCI and daily for 4 weeks.
   * Standard of care will given to both arms (group 2 and 3) and includes:

Dual Antiplatelet Therapy (DAPT), high intensity statin, anticoagulation therapy, ACEI or aldosterone antagonist depending on the ejection fraction

* All subjects will sign an informed consent statement prior to inclusion in the study.
* All subjects will be followed up for 4 weeks and blood samples will be withdrawn at baseline, 1 week, and the end of the study to test for ST2 (suppression of tumerogenicity 2) biomarker

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged >18 and < 75 years
2. Diabetic post myocardial infarction patients
3. First anterior STEMI with successful TIMI-3 flow
4. STEMI within 12 hrs of onset of chest pain
5. creatine clearance ≥60 mL/min
6. HbA1c between 6.5% and 12.0%

Exclusion Criteria:

1. Cardiogenic shock on admission
2. Multivessel disease on admission
3. Mechanical complications e.g. mitral regurge on admission
4. Life threatening arrhythmia on admission
5. Hemodynamic instability on admission
6. Diagnosis of Type 1 diabetes mellitus
7. History of bladder cancer or history of radiation therapy to the lower abdomen or pelvis at any time
8. Active urinary infection diagnosed by clinical symptoms of urgency and frequency + lab tests
9. Pregnant or breast-feeding patients
10. Active participation in another clinical study
11. AST or ALT >3x ULN or Total bilirubin >2.5 x ULN
12. CrCl < 60 ml/min (based on the Cockroft-Gault equation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Effect on ST2 (suppression of tumerogenicity 2) level in the acute phase after myocardial infarction | 4 weeks
  patients will be followed up for the whole period of the study and blood sample will be drawn at baseline and at study end to track changes in the level of ST2 (suppression of tumerogenicity 2) which is a cardiac remodeling biomarker using ELISA technique

SECONDARY OUTCOMES:
Echocardiographic changes due to intervention | 4 weeks
  patients will have their echocardiography and ejection fraction will be compared at baseline and at the end of the study to track any changes that may be caused by intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker ML, Perazella MA. SGLT2 inhibitor therapy in patients with type-2 diabetes mellitus: is acute kidney injury a concern? J Nephrol. 2020 Oct;33(5):985-994. doi: 10.1007/s40620-020-00712-5. Epub 2020 Feb 18. PMID 32067179
- [Background] Berezin AE, Berezin AA. Adverse Cardiac Remodelling after Acute Myocardial Infarction: Old and New Biomarkers. Dis Markers. 2020 Jun 12;2020:1215802. doi: 10.1155/2020/1215802. eCollection 2020. PMID 32626540
- [Background] Bolognese L, Falsini G, Schwenke C, Grotti S, Limbruno U, Liistro F, Carrera A, Angioli P, Picchi A, Ducci K, Pierli C. Impact of iso-osmolar versus low-osmolar contrast agents on contrast-induced nephropathy and tissue reperfusion in unselected patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention (from the Contrast Media and Nephrotoxicity Following Primary Angioplasty for Acute Myocardial Infarction [CONTRAST-AMI] Trial). Am J Cardiol. 2012 Jan 1;109(1):67-74. doi: 10.1016/j.amjcard.2011.08.006. Epub 2011 Sep 22. PMID 21943940
- [Background] Broch K, Andreassen AK, Ueland T, Michelsen AE, Stueflotten W, Aukrust P, Aakhus S, Gullestad L. Soluble ST2 reflects hemodynamic stress in non-ischemic heart failure. Int J Cardiol. 2015 Jan 20;179:378-84. doi: 10.1016/j.ijcard.2014.11.003. Epub 2014 Nov 5. PMID 25464491
- [Background] Brown AJM, Gandy S, McCrimmon R, Houston JG, Struthers AD, Lang CC. A randomized controlled trial of dapagliflozin on left ventricular hypertrophy in people with type two diabetes: the DAPA-LVH trial. Eur Heart J. 2020 Sep 21;41(36):3421-3432. doi: 10.1093/eurheartj/ehaa419. PMID 32578850
- [Background] Gruzdeva O, Dyleva Y, Uchasova E, Akbasheva O, Karetnikova V, Kashtalap V, Shilov A, Polikutina O, Slepynina Y, Barbarash O. Biological markers and cardiac remodelling following the myocardial infarction. Aging (Albany NY). 2019 Jun 10;11(11):3523-3535. doi: 10.18632/aging.101994. PMID 31182683
- [Background] Iwahana H, Yanagisawa K, Ito-Kosaka A, Kuroiwa K, Tago K, Komatsu N, Katashima R, Itakura M, Tominaga S. Different promoter usage and multiple transcription initiation sites of the interleukin-1 receptor-related human ST2 gene in UT-7 and TM12 cells. Eur J Biochem. 1999 Sep;264(2):397-406. doi: 10.1046/j.1432-1327.1999.00615.x. PMID 10491084
- [Background] Januzzi JL Jr, Peacock WF, Maisel AS, Chae CU, Jesse RL, Baggish AL, O'Donoghue M, Sakhuja R, Chen AA, van Kimmenade RR, Lewandrowski KB, Lloyd-Jones DM, Wu AH. Measurement of the interleukin family member ST2 in patients with acute dyspnea: results from the PRIDE (Pro-Brain Natriuretic Peptide Investigation of Dyspnea in the Emergency Department) study. J Am Coll Cardiol. 2007 Aug 14;50(7):607-13. doi: 10.1016/j.jacc.2007.05.014. Epub 2007 Jul 30. PMID 17692745
- [Background] Kokkoz C, Bilge A, Irik M, Dayangac HI, Hayran M, Akarca FK, Erdem NB, Cavus M. Prognostic value of plasma ST2 in patients with non-ST segment elevation acute coronary syndrome. Turk J Emerg Med. 2018 Feb 9;18(2):62-66. doi: 10.1016/j.tjem.2018.01.003. eCollection 2018 Jun. PMID 29922732
- [Background] Lam CSP, Chandramouli C, Ahooja V, Verma S. SGLT-2 Inhibitors in Heart Failure: Current Management, Unmet Needs, and Therapeutic Prospects. J Am Heart Assoc. 2019 Oct 15;8(20):e013389. doi: 10.1161/JAHA.119.013389. Epub 2019 Oct 12. No abstract available. PMID 31607208
- [Background] Li C, Zhang J, Xue M, Li X, Han F, Liu X, Xu L, Lu Y, Cheng Y, Li T, Yu X, Sun B, Chen L. SGLT2 inhibition with empagliflozin attenuates myocardial oxidative stress and fibrosis in diabetic mice heart. Cardiovasc Diabetol. 2019 Feb 2;18(1):15. doi: 10.1186/s12933-019-0816-2. PMID 30710997
- [Background] Ma ZG, Yuan YP, Wu HM, Zhang X, Tang QZ. Cardiac fibrosis: new insights into the pathogenesis. Int J Biol Sci. 2018 Sep 7;14(12):1645-1657. doi: 10.7150/ijbs.28103. eCollection 2018. PMID 30416379
- [Background] Mancini GB, Dahlof B, Diez J. Surrogate markers for cardiovascular disease: structural markers. Circulation. 2004 Jun 29;109(25 Suppl 1):IV22-30. doi: 10.1161/01.CIR.0000133443.77237.2f. No abstract available. PMID 15226248
- [Background] McCarthy CP, Januzzi JL Jr. Soluble ST2 in Heart Failure. Heart Fail Clin. 2018 Jan;14(1):41-48. doi: 10.1016/j.hfc.2017.08.005. PMID 29153199
- [Background] Millar NL, O'Donnell C, McInnes IB, Brint E. Wounds that heal and wounds that don't - The role of the IL-33/ST2 pathway in tissue repair and tumorigenesis. Semin Cell Dev Biol. 2017 Jan;61:41-50. doi: 10.1016/j.semcdb.2016.08.007. Epub 2016 Aug 10. PMID 27521518
- [Background] Sanada S, Hakuno D, Higgins LJ, Schreiter ER, McKenzie AN, Lee RT. IL-33 and ST2 comprise a critical biomechanically induced and cardioprotective signaling system. J Clin Invest. 2007 Jun;117(6):1538-49. doi: 10.1172/JCI30634. Epub 2007 May 10. PMID 17492053
- [Background] Santos-Gallego CG, Requena-Ibanez JA, San Antonio R, Ishikawa K, Watanabe S, Picatoste B, Flores E, Garcia-Ropero A, Sanz J, Hajjar RJ, Fuster V, Badimon JJ. Empagliflozin Ameliorates Adverse Left Ventricular Remodeling in Nondiabetic Heart Failure by Enhancing Myocardial Energetics. J Am Coll Cardiol. 2019 Apr 23;73(15):1931-1944. doi: 10.1016/j.jacc.2019.01.056. PMID 30999996
- [Background] Schmitz J, Owyang A, Oldham E, Song Y, Murphy E, McClanahan TK, Zurawski G, Moshrefi M, Qin J, Li X, Gorman DM, Bazan JF, Kastelein RA. IL-33, an interleukin-1-like cytokine that signals via the IL-1 receptor-related protein ST2 and induces T helper type 2-associated cytokines. Immunity. 2005 Nov;23(5):479-90. doi: 10.1016/j.immuni.2005.09.015. PMID 16286016
- [Background] Smith JN, Negrelli JM, Manek MB, Hawes EM, Viera AJ. Diagnosis and management of acute coronary syndrome: an evidence-based update. J Am Board Fam Med. 2015 Mar-Apr;28(2):283-93. doi: 10.3122/jabfm.2015.02.140189. PMID 25748771
- [Background] Teh PP, Vasanthakumar A, Kallies A. Development and Function of Effector Regulatory T Cells. Prog Mol Biol Transl Sci. 2015;136:155-74. doi: 10.1016/bs.pmbts.2015.08.005. Epub 2015 Sep 26. PMID 26615096
- [Background] Tominaga S. A putative protein of a growth specific cDNA from BALB/c-3T3 cells is highly similar to the extracellular portion of mouse interleukin 1 receptor. FEBS Lett. 1989 Dec 4;258(2):301-4. doi: 10.1016/0014-5793(89)81679-5. PMID 2532153
- [Background] Trajkovic V, Sweet MJ, Xu D. T1/ST2--an IL-1 receptor-like modulator of immune responses. Cytokine Growth Factor Rev. 2004 Apr-Jun;15(2-3):87-95. doi: 10.1016/j.cytogfr.2004.02.004. PMID 15110792
- [Background] Tseng CCS, Huibers MMH, van Kuik J, de Weger RA, Vink A, de Jonge N. The Interleukin-33/ST2 Pathway Is Expressed in the Failing Human Heart and Associated with Pro-fibrotic Remodeling of the Myocardium. J Cardiovasc Transl Res. 2018 Feb;11(1):15-21. doi: 10.1007/s12265-017-9775-8. Epub 2017 Dec 28. PMID 29285671
- [Background] Veeraveedu PT, Sanada S, Okuda K, Fu HY, Matsuzaki T, Araki R, Yamato M, Yasuda K, Sakata Y, Yoshimoto T, Minamino T. Ablation of IL-33 gene exacerbate myocardial remodeling in mice with heart failure induced by mechanical stress. Biochem Pharmacol. 2017 Aug 15;138:73-80. doi: 10.1016/j.bcp.2017.04.022. Epub 2017 Apr 25. PMID 28450225
- [Background] Weinberg EO, Shimpo M, De Keulenaer GW, MacGillivray C, Tominaga S, Solomon SD, Rouleau JL, Lee RT. Expression and regulation of ST2, an interleukin-1 receptor family member, in cardiomyocytes and myocardial infarction. Circulation. 2002 Dec 3;106(23):2961-6. doi: 10.1161/01.cir.0000038705.69871.d9. PMID 12460879
- [Background] Wojcik C, Warden BA. Mechanisms and Evidence for Heart Failure Benefits from SGLT2 Inhibitors. Curr Cardiol Rep. 2019 Sep 14;21(10):130. doi: 10.1007/s11886-019-1219-4. PMID 31522263